CLINICAL TRIAL: NCT01102257
Title: Clinical Trial of Essential Fatty Acids for Dry Eye Disease: Feasibility Study
Brief Title: Dry Eye Assessment and Management: Feasibility Study
Acronym: DREAM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Asbell, Penny, M.D. (Individual)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Penny Asbell, Professor, Asbell, Penny, M.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-1099; 1R34EY017626 (NIH)
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-07

CONDITIONS: Dry Eye Syndromes; Keratoconjunctivitis Sicca
Keywords: Dry Eye Disease; DED; Keratoconjunctivitis Sicca; Omega-3
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 EFA Supplement (Experimental): The total daily dose from the 5 capsules in treatment group will be 3.0 grams of omega-3 esssential fatty acid i.e Omega-3 EFA supplement comprised of:
  2000 mg EPA 1000 mg DHA
  Interventions: Drug: Omega-3 EFA Supplement
- Olive Oil (Placebo Comparator): Gel Capsule
  Interventions: Drug: Olive Oil

INTERVENTIONS:
Drug: Omega-3 EFA Supplement — The total daily dose from the 5 capsules in treatment group will be 3.0 grams of omega-3 EFAs comprised of:
  2000 mg EPA 1000 mg DHA
  Other Names: Fish oil supplements
  Arms: Omega-3 EFA Supplement
Drug: Olive Oil — Placebo group will take 5 capsules a day containing 3.0 grams of olive oil
  Arms: Olive Oil

SUMMARY:
The purpose of this study is to test a protocol investigating the efficacy of omega-3 fatty acids in treating dry eye disease. The study is termed "feasibility" because its purpose is to demonstrate an ability to execute the proposed protocol with compliance at two sites rather than generate statistically relevant data concerning the safety and efficacy of the supplement in patients with dry eye disease.

DETAILED DESCRIPTION:
Dry eye disease (DED) is a common but often inadequately treated disease of the tears and surface of the eye. It can cause poor vision and chronic pain and is more frequent with increasing age. Inflammation may be an important component of this disease. This is supported by the observation that cyclosporine, a drug that targets the immune system, is approved for and effectively treats DED. Inflammatory processes likely produce ocular surface damage and contribute to chronic DED. Because not all people with DED respond to current anti-inflammatory treatments, other immune-modulating treatments would be of value. Furthermore, despite a great deal of evidence supporting DED as an inflammatory disease, not all researchers currently agree with this classification. More data that specifically measures inflammatory responses in DED needs to be collected in a well-characterized patient population and correlated with signs and symptoms of DED in order to improve our understanding and classification of the disease.

Essential Fatty Acids (EFA) have been shown to diminish inflammatory responses in many human inflammatory diseases, and interest in the use of omega-3 and omega-6 fatty acids for disease treatment has resulted in several small studies as well as the use (and over-the-counter availability) of EFA-containing nutritional supplements, including several specifically for the treatment of DED. Despite this interest in EFA for DED, there are no strong empirical data from a well-controlled randomized controlled trial RCT supporting the use of EFA for DED. We postulate that DED is an inflammatory disease and hypothesize that EFA can mediate immune responses, thus improving DED signs, symptoms and associated measures of inflammation. The proposed three month feasibility study allows us the chance to demonstrate our ability to successfully execute our own protocol with compliance from the study patients before we begin the process of initiating a full-scale multi-center trial.

ELIGIBILITY:
Inclusion Criteria:

1. Sign and date the informed consent form approved by the IRB.
2. ≥ 18 years of age
3. Demonstrate at least 2 of the 4 following signs in the same eye at two consecutive visits (Visit 1: 7 - 21 days prior to randomization, and Visit 2: day of randomization).

   1. Conjunctival staining present ≥ 1
   2. Corneal fluorescein staining present ≥ 1
   3. Tear film break up time (TFBUT) ≤ 7 seconds
   4. Schirmer test ≤ 7 mm/5min
4. Demonstrate symptoms of dry eye disease (OSDI score of at least 22 at screening visit and at least 15 at randomization visit).
5. Use or desire to use artificial tears on average of 2 times per day in the 2 weeks preceding study entry (run in period). No newly diagnosed patients can be enrolled and if a new patient wants to participate, she/he must be put on tears and re-evaluated in 6 months.
6. Intraocular pressure (IOP) ≥ 5 mmHg and ≤ 22 mmHg in each eye.
7. Women of child-bearing potential must agree to use a reliable method of contraception during study participation, and must demonstrate a negative urine pregnancy test at screening visit.
8. Be willing/able to return for all study visits and to follow instructions from the study investigator and his/her staff.
9. Be able to swallow large, soft gelcaps

Exclusion Criteria:

1. Patients who are allergic to ingredients of the active or placebo pills (fish, olive oil).
2. Current diagnosis of ocular infection (e.g. bacterial, viral or fungal).
3. History of ocular herpetic keratitis.
4. Eye surgery (including cataract surgery) within 6 months prior to randomization.
5. Previous LASIK surgery
6. Pregnant or nursing/lactating
7. Participation in a study of an investigational drug or device within the past 30 days.
8. Recent (≤ 3 months) initiation of use of systemic corticosteroids or other immunosuppressive agent and/or is planning to change treatment during study participation
9. Cognitive or psychiatric deficit that precludes informed consent or ability to perform requirements of the investigation.
10. Contact lens wearers
11. Use of glaucoma medication or history of surgery for glaucoma.
12. Recent (≤ 3 months) insertion of punctual plugs.
13. Using punctual plugs but unwilling to commit to their use for the duration of the study.
14. Unwilling to commit to same brand of artificial tears throughout the study.
15. Current use of EPA/DHA supplements in excess of 1 gram/day.
16. Recent (≤ 6 months) initiation of use of Restasis.
17. Use of Restasis but unwilling to commit to use of Restasis for the duration of the study.
18. Discontinued use of Restasis within the last 3 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Penny Asbell, • MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Omega-3 Supplement: 5 Gel Capsules to be taken orally daily to give a total dose of 2000mg EPA and 1000 mg DHA
- Olive Oil: 5 Gel Capsules of olive oil to be taken orally daily
Period: Overall Study
Arm/Group | Omega-3 Supplement | Olive Oil
Started | 9 | 9
Completed | 7 (2 withdrew from the study d/t adverse events. 1 had shortness of breath and the other had chest pain) | 9
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Omega-3 Supplement: 5 Gel Capsules taken orally to achieve a daily dose of 2000mg EPA and 1000mg DHA
- Olive Oil: 5 Gel Capsules of olive oil taken orally daily
- Total: Total of all reporting groups
Arm/Group | Omega-3 Supplement | Olive Oil | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 3 | 3 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (14) | 57 (15) | 56 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change on Ocular Surface Disease Index (OSDI)
Time Frame: 90 +/- 14 days following initiation of drug regimen
Reporting Status: Not Posted

2. Secondary Outcome: Change on Brief Ocular Discomfort Inventory (BODI)
Time Frame: 90 +/- 14 days following initiation of drug regimen
Reporting Status: Not Posted

3. Secondary Outcome: Change on Impact of Dry Eye on Everyday Life (IDEEL)
Time Frame: 90 +/- 14 days following initiation of drug regimen
Reporting Status: Not Posted

4. Secondary Outcome: Change in Quality of Life Associated With Chronic Pain
Time Frame: 90 +/- 14 days following initiation of drug regimen
Reporting Status: Not Posted

5. Secondary Outcome: Change in the Ocular Surface
Time Frame: 90 +/- 14 days following initiation of drug regimen
Reporting Status: Not Posted

6. Secondary Outcome: Change in Schirmer's
Time Frame: 90 +/- 14 days following initiation of drug regimen
Reporting Status: Not Posted

7. Secondary Outcome: Change in Relevant Biomarkers: HLA-DR, MUC 5A, Cytokines
Time Frame: 90 +/- 14 days following initiation of drug regimen
Reporting Status: Not Posted

8. Primary Outcome: Change in REd Blood Cell(RBC) Membrane Fatty Acid(FA) Content
Time Frame: Baseline and 3 Months
Measure: Median (Inter-Quartile Range); unit: Percentage Total Fatty Acids
Arm/Group | Omega-3 Supplement | Olive Oil
Number analyzed (Participants) | 7 | 9
Percentage Total Fatty Acids
  eicosapentaenoic acid(EPA) | 1.46 [0.23 to 2.39] | 0.05 [-0.01 to 0.09]
  docosahexaenoic acid(DHA) | 1.49 [-0.36 to 1.90] | 0.25 [-0.20 to 0.36]
  Arachdinocic acid(AA) | -1.91 [-3.17 to -0.97] | -0.23 [-0.84 to -0.05]
Statistical Analysis 1: Comparison: Omega-3 Supplement vs Olive Oil; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Omega-3 Supplement | Olive Oil
Serious Adverse Events (participants affected / at risk) | 2/9 | 1/9
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Supplement (N=9) | Olive Oil (N=9)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adnexal mass due to graft verus host disease (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Omega-3 Supplement (N=4) | Olive Oil (N=2)
watery eyes (Eye disorders) | 1/1 (1) | 1/1 (1)
thirst (Nervous system disorders) | 1/1 (1) | 1/1 (1)
nausea (Nervous system disorders) | 2/2 (2) | 0/0 (0)

LIMITATIONS AND CAVEATS:
DREAM: Feasibility Study, is labeled "feasibility" because its primary end-point is to demonstrate an ability to execute the protocol rather than generate statistically relevant data on the safety and efficacy of omega-3 EFA in patients with DED.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes